CLINICAL TRIAL: NCT05501834
Title: Anxiety Surrounding Supracondylar Pin Removal in Children: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Yi-Meng Yen, Assistant Professor of Orthopedic Surgery, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00039559
Record Dates: First submitted 2022-08-02; First posted 2022-08-15 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Supracondylar Humerus Fracture; Anxiety
Keywords: Closed reduction percutaneous pinning; Supracondylar Humerus Fracture; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Both arms will receive the same Standard of Care procedures but will receive them in a different order. Patients in the control group will: 1. Go to cast room for cast removal, 2. Go to radiology for X-ray, 3. Will be seen in clinic room for pin removal. These steps are our current standard of care. An orthopedic, cast room technician bivalves and removes the top half of the patient's cast. In radiology, anteroposterior (AP) and lateral X-ray views are obtained to confirm radiographic healing. In the clinic room, a surgeon or nurse removes the pins using pin removal pliers. The order of these procedures is the current Standard of Care.
- Intervention Group (Experimental): Both arms will receive the same Standard of Care procedures but will receive them in a different order. Patients in the treatment group will: 1. Go to cast room for cast removal, 2. Have pins immediately pulled after cast removal, 3. Go to radiology for X-ray, 4. Will be seen in clinic room by provider.
  Interventions: Other: Supracondylar Pin Removal Before Imaging

INTERVENTIONS:
Other: Supracondylar Pin Removal Before Imaging — Patients in the treatment group will: 1. Go to cast room for cast removal, 2. Have pins immediately pulled after cast removal, 3. Go to radiology for X-ray, 4. Will be seen in clinic room by provider. The order of these steps differs from our current standard of care, during which patients' pins are removed following cast removal and x-ray imaging.
  Arms: Intervention Group

SUMMARY:
This study aims to determine if removing supracondylar pins immediately following cast removal and prior to X-ray decreases patient and parent/guardian anxiety compared to pin removal following cast removal and X-ray. The research team hypothesizes that patient anxiety response will be lower when pins are removed immediately following cast removal compared to our current standard of care. Secondarily, this study will determine if there is an association between patient anxiety response and their parent's/guardian's anxiety.

DETAILED DESCRIPTION:
Supracondylar humerus (SCH) fractures are one of the most common pediatric injuries. These fractures are reported as the second most common pediatric fracture, constituting about 18% of all pediatric fractures and approximately 60% of all elbow fractures. The median age of injury is between 3 and 8 years old, peaking at 5 to 6 years old. The gold standard for treating displaced SCH fractures is closed reduction and percutaneous pinning (CRPP); pins are almost always removed three to four weeks post-surgery in outpatient clinics, without anesthesia.

Many would assume that patients experience anxiety during pin removal, but no studies to our knowledge quantified a patient's physiological and behavioral response during this procedure. However, there have been many in-depth investigations of these responses during cast removal procedures, where heart rate (HR) is used as a psychological indicator of anxiety. Additionally, Merkel et al. developed the Face, Legs, Activity, Cry and Consolability (FLACC) Scale which is a valid and reliable tool to quantify pain behaviors in children. Further research showed that the FLACC Scale was also sensitive to painless procedures (i.e. intravenous insertion), and therefore, it can be considered a composite of pain and distress (anxiety).

Anxiety in the medical setting has been linked to future adverse effects for children. Previous publications have shown that patients with anxiety in the perioperative setting have increased postoperative pain, maladaptive behavior, and long-term anxiety with future medical visits. Preoperative anxiety in children also has been reported to have similar negative effects on behavior. It is plausible that an anxiety-provoking procedure, such as pin removal, would have similar effects.

The primary purpose of the first phase of this study (IRB-P00028933), which took place from 2018 to 2020, was to quantify the anxiety experienced by patients undergoing pin removal in clinic following closed reduction and percutaneous pinning (CRPP) for SCH fractures. Now that the first phase is complete, the research team is interested in taking this research another step forward to see how healthcare providers can reduce patient and parent anxiety in clinical settings. Before the first phase of this study, there were no known studies that quantified a patient's physiological and behavioral response during a postoperative pin removal procedure, as CRPP is the gold standard treatment for displaced supracondylar humerus (SCH) fractures. The findings of the primary purpose of the first phase ultimately demonstrated that all patients undergoing pin removal experience an anxiety response, therefore highlighting an area of clinical practice in need of a targeted to help decrease patient anxiety and improve patient experience.

Patients currently proceed with the following clinical flow on the day of their pin removal: (1) patients first present to the cast room for cast removal, (2) radiographs are obtained to confirm alignment and fracture stability, and (3) patients are seen by their provider in an orthopaedic clinic room for pin removal. While this process is streamlined in a busy orthopaedic clinic, it could still take up to an hour of time. After cast removal may also be the first time a patient sees the pins and this added time before pin removal could escalate anxiety. It is evident in the literature that an X-ray prior to pin removal is unnecessary, as it does not change clinical management. Anxiety in the medical setting has been linked to future adverse effects for children, such as increased postoperative pain, maladaptive behavior, and long-term anxiety with future medical visits. It is plausible that an anxiety-provoking procedure, such as pin removal, could have similar effects. Ultimately, the findings of the first phase of our study provide the groundwork for future research efforts in techniques to minimize anxiety for the pediatric patient having to undergo pin removal. Something as simple as changing the clinic flow of our current pin removal process, such as removing pins immediately following cast removal and prior to X-ray, may decrease the overall time waiting for pin removal and decrease patient anxiety.

Therefore, the primary aim of this study is to determine if removing supracondylar pins immediately following cast removal and prior to X-ray decreases patient and parent/guardian anxiety compared to pin removal following cast removal and X-ray. It is hypothesized that patient anxiety response will be lower when pins are removed immediately following cast removal compared to our current standard of care. Secondarily, this study will aim to determine if there is an association between patient anxiety response and their parent's/guardian's anxiety.

After consenting to participate in the trial, patients will be randomized to one of two treatment arms--the intervention or the control-that will be evaluated for this study. We will measure patient and parent/guardian anxiety on the day of pin removal. We plan to randomize patients into two clinical flows: standard of care clinic flow (control treatment) and change in clinic flow (new treatment).

Control Group Patients in the control group will: 1. Go to cast room for cast removal, 2. Go to radiology for X-ray, 3. Will be seen in clinic room for pin removal. These steps are our current standard of care. An orthopedic, cast room technician bivalves and removes the top half of the patient's cast. In radiology, anteroposterior (AP) and lateral X-ray views are obtained to confirm radiographic healing. In the clinic room, a surgeon or nurse removes the pins using pin removal pliers.

Intervention Group Patients in the treatment group will: 1. Go to cast room for cast removal, 2. Have pins immediately pulled after cast removal, 3. Go to radiology for X-ray, 4. Will be seen in clinic room by provider

In both groups, the study coordinator will record FLACC score and HR for patients and STAIS-5 score for parents/guardian. Training to administer the FLACC will include discussion led by the PI (Yi-Meng Yen, MD, PhD) about the 5 categories, clarification of defining characteristics for behaviors, and scoring techniques. Additionally, the study coordinator has already been trained to administer the FLACC and can also teach other study coordinators. If multiple study coordinators are used to administer the FLACC, reliability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3 to ≤8 years at time of surgery
* Supracondylar humerus fractures that are laterally pinned at Boston Children's Hospital
* Scheduled visit for pin removal at either Boston or Waltham orthopedic clinic by a study-participating physician
* English speaking

Exclusion Criteria:

* Patient diagnosed with autism

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Face, Legs, Activity, Cry and Consolability (FLACC) scale | During Treatment (Pin Removal Visit post closed reduction and percutaneous pinning)
  The Face, Legs, Activity, Cry and Consolability scale is validated in both young, non-verbal children and older, verbal children. The FLACC scale measures a patient's response to pain or distress using assessments of (1) facial expression, (2) leg movement, (3) activity, (4) extent to which they cried, and (5) extent to which they are consoled on a scale from 0 to 2 to generate a total score ranging from 0 (no pain/distress) to 10 (maximum pain/distress), with a higher score representing higher rates of anxiety and stress.
Heart rate | During Treatment (Pin Removal Visit post closed reduction and percutaneous pinning)
  Heart rate will be measured using a pulse oximetry heart rate monitor. We plan to use heart rate as a physiological correlate to the FLACC scale. For the purposes of this study, we will define an anxiety response as any patient who scores greater than 0 on the FLACC or achieves a HR in excess of the upper 95% normative limits for their age, sex and race (where applicable).

SECONDARY OUTCOMES:
Face, Legs, Activity, Cry and Consolability (FLACC) scale | During Treatment (Pin Removal Visit post closed reduction and percutaneous pinning)
  The Face, Legs, Activity, Cry and Consolability scale is validated in both young, non-verbal children and older, verbal children. The FLACC scale measures a patient's response to pain or distress using assessments of (1) facial expression, (2) leg movement, (3) activity, (4) extent to which they cried, and (5) extent to which they are consoled on a scale from 0 to 2 to generate a total score ranging from 0 (no pain/distress) to 10 (maximum pain/distress), with a higher score representing higher rates of anxiety and stress.
Heart rate | During Treatment (Pin Removal Visit post closed reduction and percutaneous pinning)
  Heart rate will be measured using a pulse oximetry heart rate monitor. We plan to use heart rate as a physiological correlate to the FLACC scale. For the purposes of this study, we will define an anxiety response as any patient who scores greater than 0 on the FLACC or achieves a HR in excess of the upper 95% normative limits for their age, sex and race (where applicable).
Spielberger State-Trait Anxiety Inventory (STAI-5) | During Treatment (Pin Removal Visit post closed reduction and percutaneous pinning)
  The Spielberger State-Trait Anxiety Inventory (STAI-5) has been widely used to measure the state and trait components of anxiety. The STAI has been shown to have excellent psychometric properties with good reliability and validity. The questionnaire can measure anxiety both in healthy and in clinical populations, with those scoring higher on STAI scales indicating to be more prone to experience anxiety. We plan to use this to measure the parent/guardian anxiety response to patient pin removal.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Meng Yen, MD, PhD, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: No